CLINICAL TRIAL: NCT03330223
Title: Effect of Haemodialysis on the Efficacy of Antiplatelet Agents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 008
Record Dates: First submitted 2017-09-27; First posted 2017-11-06 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-09

CONDITIONS: Renal Failure; Coronary Artery Disease; Hemolysis
MeSH Terms: conditions — Renal Insufficiency; Coronary Artery Disease; Hemolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clopidogrel: clopidogrel 75mg qd;aspirin 100mg qd, n=30
  Interventions: Device: Clopidogrel group;Ticagrelor group
- Ticagrelor: ticagrelor 90mg bid; aspirin 100mg qd, n=30
  Interventions: Device: Clopidogrel group;Ticagrelor group

INTERVENTIONS:
Device: Clopidogrel group;Ticagrelor group — A total of 60 patients with ESRD and under dual-antiplatelet treatmen for at least 5 days will be enrolled and divided into the Clopidogrel group (clopidogrel 75mg qd;aspirin 100mg qd, n=30) and the Ticagrelor group (ticagrelor 90mg bid; aspirin 100mg qd, n=30). All included patients will receive haemodialysis by two different types of dialysis membrane.Platelet aggregation of venous blood from all patients will be detected by LTA and VerifyNow immediately before and after haemodialysis.

SUMMARY:
The main purpose of our study is to investigate whether haemodialysis itself affects the efficacy of antiplatelet drugs and the effects of two different types of dialysis membranes (polysulfone membranes and polyamide membranes) on antiplatelet efficacy. A total of 60 patients with ESRD and under dual-antiplatelet treatmen for at least 5 days will be enrolled and divided into the Clopidogrel group (clopidogrel 75mg qd;aspirin 100mg qd, n=30) and the Ticagrelor group (ticagrelor 90mg bid; aspirin 100mg qd, n=30). All included patients will receive haemodialysis by two different types of dialysis membrane.Platelet aggregation of venous blood from all patients will be detected by LTA and VerifyNow immediately before and after two times of haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of coronary heart disease including stable angina, unstable angina, acute myocardial infarction
* taking dual antiplatelet drugs (clopidogrel 75mg qd + aspirin 100mg qd or ticagrelor 90 mg,bid + aspirin 100 mg,qd) at least 5 days
* haemodialysis patients
* sign informed consent

Exclusion Criteria:

* platelet count>450 × 10 9 /L or <100 × 10 9 /L
* using IIb / IIIa inhibitor drugs within 10days
* taking nonsteroidal anti-inflammatory drugs other than aspirin
* hemorrhagic disease
* allergic to aspirin, ticagrelor or clopidogrel
* other factors may affect the results of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiovascular events account for about 50% of all-cause mortality in patients with end-stage renal disease(ESRD), and about 20% of cardiac death events are caused by acute coronary syndromes(ACS).Over the past decade, the number of percutaneous coronary intervention (PCI) in patients with ESRD has increased by nearly 50%. Aspirin, clopidogrel and ticagrelor are the most widely used antiplatelet agents in ACS patients after PCI.Little is known about whether hemodialysis can affect the efficacy of antiplatelet agents or not.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
using light transmittance aggregometer to detect whether haemodialysis can affect the efficacy of antiplatelet agents | collecting blood within 10 miuntes before and after haemodialysis;detecting them within 2 hours
  intravenous blood collection with anticoagulant tube before and after haemodialysis respectively ；using light transmittance aggregometer to detect adenosine diphosphate induced platelet aggregation rate and arachidonic acid induced platelet aggregation rate within two hours after blood collection;;compare the outcome of light transmittance aggregometer with VerifyNow

SECONDARY OUTCOMES:
using VerifyNow to detect whether haemodialysis can affect the efficacy of antiplatelet agents | collecting blood within 10 miuntes before and after haemodialysis;detecting them within 2 hours
  intravenous blood collection with VeryfiNow to detect the platelet reaction unit before and after haemodialysis respectively

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ye Z, Wang Q, Ullah I, Lin Q, Wu T, Yang M, Fan Y, Dong Z, Wang T, Teng J, Hua R, Tang Y, Li Y, Gong X, Yuan L, Tao Z, Li C. Impact of hemodialysis on efficacies of the antiplatelet agents in coronary artery disease patients complicated with end-stage renal disease. J Thromb Thrombolysis. 2024 Apr;57(4):558-565. doi: 10.1007/s11239-023-02924-5. Epub 2024 Feb 23. PMID 38393676